CLINICAL TRIAL: NCT03344783
Title: The Effects of Early Life Polyunsaturated Fatty Acids and Ruminant Trans Fatty Acids on Allergic Diseases: A Systematic Review and Meta-analysis
Brief Title: The Effects of Early Life PUFA and R-TFA on AD: A Systematic Review and Meta-analysis
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Cai, Principal Investigator, Sun Yat-sen University
Other Study IDs: Weijia,Wu
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Allergic Disorder
MeSH Terms: conditions — Hypersensitivity | interventions — Fatty Acids, Unsaturated

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mother-children pairs
  Interventions: Other: PUFA and R-TFA

INTERVENTIONS:
Other: PUFA and R-TFA — PUFA and R-TFA exposure were assessed mainly from maternal dietary, blood sample or breast milk. Exposure period was restricted to early life. Dietary PUFA and R-TFA were measured by food-frequency questionnaire (FFQ) or diet history questionnaire (DHQ). The profile of PUFA and R-TFA in the blood sample and breast milk were examined by using gas chromatography

SUMMARY:
The purpose of this study is to evaluate whether early life natural exposure to fatty acid affects the AD risk.

DETAILED DESCRIPTION:
The prevalence of Allergic Diseases (AD) is rising dramatically worldwide especially in more industrialized countries during the past two decades, representing a substantial disease burden of individuals and health service cost. Early life nutritional exposures could modify the gene expression and susceptibility of allergic diseases (AD), yet the effects of early life polyunsaturated fatty acids (PUFA) and ruminant trans fatty acids (R-TFA) on AD remain unclear.Therefore,the investigators performed the meta-analysis and systematic review to evaluate whether early life natural exposure to PUFA and R-TFA affects the AD risk.

ELIGIBILITY:
Inclusion Criteria:

* Studies needed to provide endpoints of AD, and risk estimates [odds risk (OR), relative risk (RR) or hazard ratio (HR)] for PUFA or R-TFA as the exposure. We included English language articles only, while scanned titles /abstracts of non-English language articles to evaluate agreement with the results published in English.

Exclusion Criteria:

* Studies were excluded if they didn't report the profile of PUFA or R-TFA, or if they targeted participants with medical condition.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Among these studies, most of them were performed in Europe. The sample size ranged from 65 to 4,976, with a median sample size of 708. One study included only boys, while the others included both sexes. Mother's mean age ranged from 27.5 to 38.7 years.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Eczema were determined by using the validated International Study of Asthma and Allergic in Children (ISAAC) questionnaire or doctors' diagnosis. | From date of inclusion of pregnant women cohort until the date of eczema' diagnosis in children,follow-up time up to 18 years
  Parental reported questions adapted from the International Study on Asthma and Allergy in Childhood (ISAAC) provided information on eczema.Researchers combined questions into current eczema (no, yes).
Wheeze were determined by using the validated International Study of Asthma and Allergic in Children (ISAAC) questionnaire or doctors' diagnosis. | From date of inclusion of pregnant women cohort until the date of wheeze' diagnosis in children,follow-up time up to 18 years
  Parental reported questions adapted from the International Study on Asthma and Allergy in Childhood (ISAAC) provided information on wheeze.Researchers combined questions into current wheeze (no, yes).
Asthma were determined by using the validated International Study of Asthma and Allergic in Children (ISAAC) questionnaire or doctors' diagnosis. | From date of inclusion of pregnant women cohort until the date of asthma' diagnosis in children,follow-up time up to 18 years
  Parental reported questions adapted from the International Study on Asthma and Allergy in Childhood (ISAAC) provided information on asthma.Researchers combined questions into current asthma (no, yes).
Allergic rhinitis were determined by using the validated International Study of Asthma and Allergic in Children (ISAAC) questionnaire or doctors' diagnosis. | From date of inclusion of pregnant women cohort until the date of allergic rhinitis' diagnosis in children,follow-up time up to 18 years
  Parental reported questions adapted from the International Study on Asthma and Allergy in Childhood (ISAAC) provided information on allergic rhinitis.Researchers combined questions into current allergic rhinitis (no, yes).
Sensitization were determined by IgE test. | From date of inclusion of pregnant women cohort until the date of sensitization' diagnosis in children,follow-up time up to 18 years
  A child was considered sensitized if the IgE level for at least one of the seven allergens was ≥0.35 kUA/l, and nonsensitized if IgE level for all seven allergens was <0.35 kUA/l.

CONTACTS AND LOCATIONS:
Overall Officials: Li Cai, PhD, Study Chair — Sun Yat-sen University
Locations (1):
- Weijia, Wu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Best KP, Gold M, Kennedy D, Martin J, Makrides M. Omega-3 long-chain PUFA intake during pregnancy and allergic disease outcomes in the offspring: a systematic review and meta-analysis of observational studies and randomized controlled trials. Am J Clin Nutr. 2016 Jan;103(1):128-43. doi: 10.3945/ajcn.115.111104. Epub 2015 Dec 16. PMID 26675770
- [Background] Anandan C, Nurmatov U, Sheikh A. Omega 3 and 6 oils for primary prevention of allergic disease: systematic review and meta-analysis. Allergy. 2009 Jun;64(6):840-8. doi: 10.1111/j.1398-9995.2009.02042.x. Epub 2009 Apr 7. PMID 19392990
- [Background] Wu WF, Wan KS, Wang SJ, Yang W, Liu WL. Prevalence, severity, and time trends of allergic conditions in 6-to-7-year-old schoolchildren in Taipei. J Investig Allergol Clin Immunol. 2011;21(7):556-62. PMID 22312941